CLINICAL TRIAL: NCT03264794
Title: Evaluation of the Efficacy of Domestic Gefitinib Tablets in the Treatment of Locally Advanced or Metastatic Non-small Cell Lung Cancer Patients Using a Multicenter, Randomized, Positive Drug Gefitinib Pharmacodynamics and Pharmacodynamics
Brief Title: the Clinical Trial of Gefitinib(Non - Small Cell Lung Cancer)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Famous Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTTQ-20161017
Record Dates: First submitted 2017-07-03; First posted 2017-08-29 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-01

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- trial group (Experimental): Gefitinib tablets (CTTQ），First medication.From the 8th day of the experiment, treated with Gefitinib Tab（CTTQ）
  Interventions: Drug: Gefitinib Tab （CTTQ），First medication；Gefitinib Tab （CTTQ），From the 8th day of trial; Drug: Gefitinib Tab 250 MG（CTTQ），From the 8th day of trial.
- control group (Active Comparator): Gefitinib tablets (Yi Ruisha），First medication.From the 8th day of the experiment, treated with Gefitinib Tab（CTTQ）
  Interventions: Drug: Gefitinib tablets (Yi Ruisha），First medication; Drug: Gefitinib Tab 250 MG（CTTQ），From the 8th day of trial.

INTERVENTIONS:
Drug: Gefitinib Tab （CTTQ），First medication；Gefitinib Tab （CTTQ），From the 8th day of trial — Gefitinib Tab （CTTQ），First medication,250mg；
  Arms: trial group
Drug: Gefitinib tablets (Yi Ruisha），First medication — Gefitinib tablets (Yi Ruisha），First medication,250mg；
  Arms: control group
Drug: Gefitinib Tab 250 MG（CTTQ），From the 8th day of trial. — From the 8th day of the experiment, two groups of subjects were treated with Gefitinib（CTTQ）

SUMMARY:
1. Gefitinib CTTQ production gefitinib and erlotinib sheet AstraZeneca imatinib sheet (trade name: Iressa ®) comparison, human pharmacokinetics and relative bioavailability of comparative studies which examine people in vivo pharmacokinetic behavior, provide the basis for clinical use.
2. Evaluation CTTQ gefitinib imatinib sheet production efficacy and safety of Chinese patients with locally advanced or metastatic non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients volunteered to participate in this study, signed informed consent;
2. ≥18 years old; ECOG PS score: 0 ~ 1; expected survival period of more than 3 months;
3. patients with locally advanced or metastatic non-small cell lung cancer diagnosed by histology or cytology, who can not receive radical surgery or radiotherapy; patients with measurable lesions(according to RECIST criteria);
4. Detection of EGFR-positive exon 19 deletion or exon 21 (L858R) mutation was performed by providing a detectable specimen (tissue or cancerous pleural effusion) prior to enrollment;
5. The main organ function within 7 days before treatment, meet the following criteria:

(1) blood routine examination criteria (14 days without blood transfusion): A) hemoglobin≥ 90g / L; B) neutrophil absolute ≥ 1.5 × 109 / L; C) platelet ≥80 × 109 / L (2) biochemical tests to meet the following criteria: A) total bilirubin ≤ 1.5 times the upper limit of normal (ULN); B) alanine aminotransferase and aspartate aminotransferase AST ≤ 2.5ULN, such as liver metastasis, ALT and AST ≤ 5ULN; C) serum creatinine ≤ 1.5ULN or creatinine clearance ≥ 60ml / min; (3) Doppler ultrasound evaluation: left ventricular ejection fraction (LVEF) ≥ normal low (50%).

6.Women of childbearing age should agree that contraceptive measures (such as intrauterine devices, birth control pills or condoms) must be used within the study period and within 6 months after the end of the study; serum or urine pregnancy test is negative within 7 days prior to enrollment, And must be non-lactating patients; men should agree to patients who have contraceptive use during the study period and six months after the end of the study period.

Exclusion Criteria:

1. patients who have previously used EGFR-TKI drugs;
2. small cell lung cancer (including small cell carcinoma and non-small cell carcinoma mixed lung cancer);
3. central type, with empty lung squamous cell carcinoma, or with non-small cell lung cancer with hemoptysis (> 50 ml / day) 4.5 years or at the same time with other malignancies, cured cervical carcinoma in situ, non-melanoma skin cancer and superficial bladder tumor except [Ta (non-invasive tumor), Tis (carcinoma in situ ) And T1 (tumor infiltrating basement membrane)];

5.Whole-body antitumor therapy was planned within 4 weeks prior to randomization or during the course of this study, including cytotoxic therapy, signal transduction inhibitors, immunotherapy (or use of mitogen at 6 weeks prior to administration of the test drug) C); 6.patients with symptomatic or unstable brain metastases; 7.patients with any severe and / or uncontrolled disease, including: A) cirrhosis, acute or active hepatitis; B) history of immunodeficiency, including HIV-positive or other acquired, congenital immunodeficiency disease, or history of organ transplantation; C) patients with seizures and who need treatment; 8.active or uncontrollable serious infection (≥CTC AE Level 2 infection); 9.with a history of mental illness and can not quit or have mental disorders; 10.participated in other anti-tumor drug clinical trials within four weeks; 11.According to the judge's judgment, there is an impact on the absorption of oral drugs or serious harm to the safety of patients is not suitable for participation in the study of the situation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Gefitinib plasma concentration | 0hour before administration and 1, 2, 3, 4, 5, 6, 7, 8,9,13,24,48,72,120,168 16 hour time points after administration
  After the use of gefitinib to reach the highest plasma concentration
Tmax time | 0hour before administration and 1, 2, 3, 4, 5, 6, 7, 8,9,13,24,48,72,120,168 16 hour time points after administration
  Taking the time required for the concentration of gefitinib to reach the peak
AUC0-t | 0hour before administration and 1, 2, 3, 4, 5, 6, 7, 8,9,13,24,48,72,120,168 16 hour time points after administration
  The area between the axis of the coordinate and the time drug concentration curve
t 1/2 | 0hour before administration and 1, 2, 3, 4, 5, 6, 7, 8,9,13,24,48,72,120,168 16 hour time points after administration
  The time required for gefitinib to decrease by half the highest concentration in plasma
F | 0hour before administration and 1, 2, 3, 4, 5, 6, 7, 8,9,13,24,48,72,120,168 16 hour time points after administration
  Gefitinib absorbs the relative amount of blood into the cycle

IPD SHARING:
Plan to Share IPD: Undecided